CLINICAL TRIAL: NCT00114205
Title: Phase I Trial of Intrapleural Docetaxel Administered Via an Implantable Catheter in Subjects With a Malignant Pleural Effusion
Brief Title: Surgery and Intrapleural Docetaxel in Treating Patients With Malignant Pleural Effusion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000430930; UVACC-HIC-10722; UVACC-29303
Record Dates: First submitted 2005-06-13; First posted 2005-06-14 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2006-08

CONDITIONS: Metastatic Cancer
Keywords: malignant pleural effusion
MeSH Terms: conditions — Neoplasm Metastasis; Pleural Effusion, Malignant | interventions — Docetaxel

INTERVENTIONS:
Drug: docetaxel
Procedure: therapeutic thoracoscopy

SUMMARY:
RATIONALE: Giving drugs, such as docetaxel, directly into the pleura after surgery to drain the pleural effusion may help keep fluid from building up again.

PURPOSE: This phase I trial is studying the side effects, best way to give, and best dose of intrapleural docetaxel given after surgery in patients with malignant pleural effusion.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of intrapleural docetaxel in patients with malignant pleural effusion.

Secondary

* Determine the toxicity profile of this drug in these patients.
* Determine the pharmacokinetics of this drug in plasma and pleural fluid from these patients.
* Determine the response in patients treated with this drug.

OUTLINE: This is a dose-escalation study.

Patients undergo thorascopic surgery to drain the malignant pleural effusion. An intrapleural catheter (Pleurx catheter) is then inserted for subsequent docetaxel instillation. Approximately 24 hours after surgery, patients receive docetaxel intrapleurally over 3 minutes via the Pleurx catheter. The Pleurx catheter is then clamped for 4 hours and the patient is placed in several different positions to ensure uniform distribution of docetaxel throughout the pleural cavity.

Cohorts of 3-6 patients receive escalating doses of intrapleural docetaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

After completion of study treatment, patients are followed at weeks 1 and 3 and then monthly thereafter.

PROJECTED ACCRUAL: Approximately 8-24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed malignant pleural effusion (MPE)

  * Symptomatic disease
* Candidate for thoracoscopic surgery for treatment of MPE

  * No known or suspected ipsilateral pleurodesis that would preclude surgery
* No bilateral MPEs
* No progressive extrapleural disease that is untreatable and/or resistant to systemic treatment

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8.0 g/dL

Hepatic

* ALT and/or AST ≤ 1.5 times upper limit of normal (ULN) (if alkaline phosphatase normal) OR
* Alkaline phosphatase ≤ 2.5 times ULN (if ALT and/or AST normal)
* Bilirubin normal
* INR ≤ 1.5

Renal

* Creatinine ≤ 1.8 mg/dL

Other

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 1 month after completion of study treatment
* No history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
* No peripheral neuropathy > grade 1

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No concurrent systemic chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2003-07

PRIMARY OUTCOMES:
Maximum tolerated dose by adverse event evaluation 1 month after treatment

SECONDARY OUTCOMES:
Pharmacokinetics by serum and pleural fluid analyses through 1 month
Clinical response by chest x-ray response and survival

CONTACTS AND LOCATIONS:
Overall Officials: David R. Jones, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Cancer Center, Charlottesville, Virginia, United States